CLINICAL TRIAL: NCT03478020
Title: Open-Label, Fixed-Sequence 3-Period Study to Determine the Effects of Repeated Oral Dosing of AQX-1125 on the Pharamacokinetics, Safety and Tolerability of a Combination Oral Contraceptive in Healthy Female Subjects
Brief Title: Oral AQX-1125 and Combination Oral Contraceptive Drug-Drug Interaction Study
Acronym: DDI-COC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aquinox Pharmaceuticals (Canada) Inc. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AQX-1125-104
Record Dates: First submitted 2018-03-19; First posted 2018-03-27 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — 4-(4-(aminomethyl)-7a-methyl-1-methylideneoctahydro-1H-inden-5-yl)-3-(hydroxymethyl)-4-methylcyclohexan-1-ol; Contraceptives, Oral, Combined

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pre-Treatment, Treatment Cycles A & B (Experimental): Pre-Treatment: Two cycles of a combined oral contraceptive (COC) taken orally once daily for 21 days followed by 7 COC-free days.
  Treatment Period A: COC containing taken orally once daily for 21 days followed by 7 COC-free days.
  Treatment Period B: COC taken orally once daily for 21 days, with once daily oral 200 mg AQX-1125 (2 x 100 mg tablets) co-administered from Day 13 to 21, followed by 7 COC-free days
  Interventions: Drug: AQX-1125; Drug: Combined Oral Contraceptive

INTERVENTIONS:
Drug: AQX-1125 — Investigational Drug
Drug: Combined Oral Contraceptive — COC containing 100 ug Levonorgestrel (LNG) and 20 ug Ethinyl Estradiol (EE)

SUMMARY:
This is an open-label, fixed sequence, 4 cycle, drug-drug interaction (DDI) study of AQX-1125 in healthy female subjects on combination oral contraceptives (COC).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-45 years, inclusive, at time of signing Informed Consent
* Adult females of child bearing potential, who are non-pregnant and non-lactating, and must agree to use adequate additional contraception from the start of Treatment Period A until 90 days after the last dose of AQX-1125
* BMI 18.0 - 35.0 kg/m2
* Good physical and mental health based on medical history, physical examination, clinical laboratory, ECG and vital signs, as judged by the investigator

Exclusion Criteria:

* Previous participation in the current study
* Any clinically significant history of breakthrough bleeding
* Using tobacco or other nicotine containing products within 12 months prior to the first study-specific COC-cycle intake
* History of alcohol abuse or drug addiction
* Positive drug and alcohol screen at screening and (each) admission to the clinical research center
* Average intake of more than 24 units of alcohol per week
* Positive screen for hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV) antibodies or anti-human immunodeficiency virus (HIV) 1 and 2 antibodies
* Participation in a drug study within 30 days prior to screening. Participation in more than 2 other drug studies in the 10 months prior to (the first) drug administration in the current study
* Donation or loss of more than 100 mL of blood within 60 days prior to the start of Treatment Period A, on Day 1. Donation or loss of more than 1.0 liters of blood in the 10 months prior to the start of Treatment Period A, on Day 1
* Significant and/or acute illness within 5 days prior to Day 1 in Treatment Period A, that may impact safety assessments, in the opinion of the investigator
* Unsuitable veins for blood sampling

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pre-Menopausal Female Subjects
Enrollment: 32 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-04-05 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of COC taken with AQX-1125 | 8 Weeks (from start of treatment period A to completion of treatment period B)
  To assess the effect of multiple doses of 200 mg AQX-1125 once daily (qd) on the pharmacokinetics (PK) of the COC
Time to attain maximum observed plasma concentration (tmax) of COC taken with AQX-1125 | 8 Weeks (from start of treatment period A to completion of treatment period B)
  To assess the effect of multiple doses of 200 mg AQX-1125 once daily (qd) on the pharmacokinetics (PK) of the COC
Area under the plasma concentration-time curve up to 24 hours (AUC0-24) of COC taken with AQX-1125 | 8 Weeks (from start of treatment period A to completion of treatment period B)
  To assess the effect of multiple doses of 200 mg AQX-1125 once daily (qd) on the pharmacokinetics (PK) of the COC
Terminal elimination rate constant (Kel) of COC taken with AQX-1125 | 8 Weeks (from start of treatment period A to completion of treatment period B)
  To assess the effect of multiple doses of 200 mg AQX-1125 once daily (qd) on the pharmacokinetics (PK) of the COC
Terminal elimination half-life (t1/2) of COC taken with AQX-1125 | 8 Weeks (from start of treatment period A to completion of treatment period B)
  To assess the effect of multiple doses of 200 mg AQX-1125 once daily (qd) on the pharmacokinetics (PK) of the COC

SECONDARY OUTCOMES:
Safety and tolerability of AQX-1125 200 mg qd administered with the COC | 16 weeks (from start of pre-treatment cycle 1 to completion of treatment period B)
  Safety and tolerability will be assessed by the severity and frequency of adverse events, which will include any abnormal clinically significant vital signs, laboratory tests, electrocardiogram and physical examination findings
Maximum observed plasma concentration (Cmax) of AQX-1125 taken with COC | 8 Weeks (from start of treatment period A to completion of treatment period B)
  To assess the PK of 200 mg AQX-1125 qd when given together with the COC
Time to attain maximum observed plasma concentration (tmax) of AQX-1125 taken with COC | 8 Weeks (from start of treatment period A to completion of treatment period B)
  To assess the PK of 200 mg AQX-1125 qd when given together with the COC
Area under the plasma concentration-time curve up to 24 hours (AUC0-24) of AQX-1125 taken with COC | 8 Weeks (from start of treatment period A to completion of treatment period B)
  To assess the PK of 200 mg AQX-1125 qd when given together with the COC
Terminal elimination rate constant (Kel) of AQX-1125 taken with COC | 8 Weeks (from start of treatment period A to completion of treatment period B)
  To assess the PK of 200 mg AQX-1125 qd when given together with the COC
Terminal elimination half-life (t1/2) of AQX-1125 taken with COC | 8 Weeks (from start of treatment period A to completion of treatment period B)
  To assess the PK of 200 mg AQX-1125 qd when given together with the COC

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen van de Wetering, MD, Principal Investigator — PRA Health Sciences
Locations (1):
- PRA Health Sciences - Early Development Serices, Groningen, Netherlands